CLINICAL TRIAL: NCT05546762
Title: IrRigation of the INfected Pleural Space With antiSEptic Solution (RINSE) - a Proof of Concept Study
Brief Title: Trial of Antiseptic Irrigation for Pleural Infection
Acronym: RINSE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Maged Hassan, Principal investigator, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02/24/09/2022
Record Dates: First submitted 2022-09-11; First posted 2022-09-21 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Empyema, Pleural
MeSH Terms: conditions — Empyema, Pleural | interventions — Saline Solution

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Antiseptic irrigation arm (Experimental): 250 ml solution of 2% povidone-iodine (i.e. 50 ml betadine in 200 ml saline) will be attached to the chest tube via a giving set and a 3-way tap and irrigated into the pleural space with gravity. The chest tube will be clamped for 10-20 minutes after irrigation and then will be unclamped and left to drain freely. The first dose will be applied 24-48 hours after tube insertion. This will be repeated every 12 hours for a total of four to six applications.
  Interventions: Drug: Povidone-iodine solution
- Saline irrigation arm (Active Comparator): 250 ml solution of normal saline will be attached to the chest tube via a giving set and a 3-way tap and irrigated into the pleural space with gravity. The chest tube will be clamped for 10-20 minutes after irrigation and then will be unclamped and left to drain freely. The first dose will be applied 24-48 hours after tube insertion. This will be repeated every 12 hours for a total of four to six applications.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Povidone-iodine solution — Pleural irrigation with 2% povidone iodine
  Arms: Antiseptic irrigation arm
Drug: Normal saline — Pleural irrigation with normal saline
  Arms: Saline irrigation arm

SUMMARY:
Pleural antiseptic irrigation (PAI) is used in conjunction with open drainage for treating adults with chronic post-thoracotomy empyema. The antiseptic povidone-iodine can safely be instilled into the pleural cavity for the purpose of pleurodesis and has recently been described for pleural irrigation in the acute management of paediatric pleural infection with good outcomes. A recent case report demonstrated the safe use of povidone-iodine pleural irrigation in a patient with complex pleural empyema with successful medical management. In a previous pilot study, antiseptic irrigation led to less referral to surgery and shorter length of hospital stay in comparison to no irrigation.

This study aims to investigate the effect of antiseptic pleural irrigation (using povidone iodine) on the inflammatory response in adults patients with pleural infection in comparison to irrigation with normal saline alone. A reduction in the systemic inflammatory response can be inferred to correlate with reduction in the infection burden in the pleural space.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 year-old or more)
* Pleural infection diagnosed by: the presence of pus in the pleural space, OR any of the following in the setting of acute lower-respiratory tract infection symptoms: pleural fluid PH<7.2 or pleural fluid glucose <40 mg/dL, positive gram stain or culture from pleural fluid
* Predominantly unilocular pleural collection treated with chest tube drainage
* Acute response at presentation as evidenced by fever (>37.80C) and/or blood leucocytosis (>11X103/mm3) and/or high serum C-reactive protein, CRP (>50 mg/L)

Exclusion Criteria:

* Known or suspected thyroid disease
* Allergy to iodine
* Persistent large collection on follow-up imaging 24-48 post tube insertion that is deemed to require additional interventions (e.g., another drainage procedure, intrapleural fibrinolytic)
* Evidence or suspicion of broncho-pleural fistula (suspected when there is air-fluid level without previous intervention, or if the participant is coughing large volume of purulent sputum that is physically similar to drained pleural fluid)
* Tuberculous, post-operative or post-haemothorax pleural infections

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-09-19 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Percentage change in inflammatory markers before and after irrigation | Initial levels to be measured 12 to 48 hours post tube insertion and follow up levels 12 to 24 hours post last dose of irrigation
  The percentage by which inflammatory marker (CRP and/or procalcitonin) decrease after completing all irrigations in comparison to the pre-irrigation inflammatory markers level

SECONDARY OUTCOMES:
Time in days to chest tube removal | At the time of chest tube removal (up to 6 weeks)
  The time in days from the first irrigation to the chest tube removal
Total length of hospital stay in days | At the point of deciding a patient is medically fit for discharge (assessed up to 6 weeks)
  Duration of hospital stay from admission until a patient is declared medically fit for discharge
Percentage of radiological clearance between baseline and discharge chest X-rays | baseline and discharge (up to week 6)
  Percentage of radiological clearance of pleural abnormalities between baseline and discharge chest X-rays using a computer software
Incidence of medical treatment failure | At discharge from the hospital or referral to another department (assessed up to week 6)
  Number of patients who fail medical treatment (referral to surgery, further pleural procedures or death)
Incidence of adverse events | Adverse events will be recognised if they appear within 6 hours of a given irrigation procedure
  Number of patients with different types of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
These spreadsheet with individual participant data will be stored after trial conclusion with the principal investigator and will be accessible to other members of the study team. Request to access study data by other researchers will be expected via email and access will be granted by the principal investigator if the request is deemed reasonable.
Time Frame: Data will be available for a minimum of five years after study conclusion
Access Criteria: Request for access will be granted when reasonable reasons for request are given

REFERENCES:
- [Background] Cargill TN, Hassan M, Corcoran JP, Harriss E, Asciak R, Mercer RM, McCracken DJ, Bedawi EO, Rahman NM. A systematic review of comorbidities and outcomes of adult patients with pleural infection. Eur Respir J. 2019 Oct 1;54(3):1900541. doi: 10.1183/13993003.00541-2019. Print 2019 Sep. PMID 31391221
- [Background] Sogaard M, Nielsen RB, Norgaard M, Kornum JB, Schonheyder HC, Thomsen RW. Incidence, length of stay, and prognosis of hospitalized patients with pleural empyema: a 15-year Danish nationwide cohort study. Chest. 2014 Jan;145(1):189-192. doi: 10.1378/chest.13-1912. No abstract available. PMID 24394842
- [Background] Mummadi SR, Stoller JK, Lopez R, Kailasam K, Gillespie CT, Hahn PY. Epidemiology of Adult Pleural Disease in the United States. Chest. 2021 Oct;160(4):1534-1551. doi: 10.1016/j.chest.2021.05.026. Epub 2021 May 20. PMID 34023322
- [Background] Hooper CE, Edey AJ, Wallis A, Clive AO, Morley A, White P, Medford AR, Harvey JE, Darby M, Zahan-Evans N, Maskell NA. Pleural irrigation trial (PIT): a randomised controlled trial of pleural irrigation with normal saline versus standard care in patients with pleural infection. Eur Respir J. 2015 Aug;46(2):456-63. doi: 10.1183/09031936.00147214. Epub 2015 May 28. PMID 26022948
- [Background] Muthu V, Dhooria S, Sehgal IS, Prasad KT, Aggarwal AN, Agarwal R. Iodopovidone pleurodesis for malignant pleural effusions: an updated systematic review and meta-analysis. Support Care Cancer. 2021 Aug;29(8):4733-4742. doi: 10.1007/s00520-021-06004-3. Epub 2021 Jan 30. PMID 33515303
- [Background] Elhoffy A, Amin A, Sadaka AS, Hassan M. Management of a complex thoracic infection, one compartment at a time. Thorax. 2022 Apr;77(4):417-419. doi: 10.1136/thoraxjnl-2021-218475. Epub 2022 Jan 17. No abstract available. PMID 35039443